CLINICAL TRIAL: NCT05542472
Title: The Effect on Caregivers of a Family Support Program Based on a Nurse-Led Case Management Model
Brief Title: The Effect on Caregivers of a Family Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, fatma tanrıkulu, Principal Investigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16214662/050.0104/127
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Caregiver Burnout
Keywords: caregiver; case management; nurse-led
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention will perform on the caregivers in the control group. The patients will continue to receive care under public services.
- Interventional group (Experimental): A Family Support Program Based on the Nurse-Led Case Management Model will create for the caregivers in the intervention group. The nurse-led case management model is made up of five basic nursing activities.
  First Nursing Activity: Determining individuals who can benefit from the case management model Second Nursing Activity: Establishing individuals' problems and care needs Third Nursing Activity: Planning nursing activities to meet the determined needs Fourth Nursing Activity: Implementing nursing activities Fifth Nursing Activity: Regular review, monitoring and assessment of nursing activities
  Interventions: Other: Family Support Program Based on a Nurse-Led Case Management Model

INTERVENTIONS:
Other: Family Support Program Based on a Nurse-Led Case Management Model — A Family Support Program Based on the Nurse-Led Case Management Model create for the care givers in the intervention group. Case management is the process of planning an individual's care, coordinating it, managing it, implementing it and reviewing it. The aim in case management is to improve a person's quality of life by coordinating health care services and providing these services at a reasonable cost and in a productive way. The use of case management requires the cooperation of professionals from many different disciplines. Therefore, in areas where case management is applied, the case manager coordinates an individual's or patient's care by enabling this cooperation. In this way, in areas where health services are provided, the case manager may be a doctor, a nurse, a physiotherapist, a social services expert, or a speech therapist.
  Arms: Interventional group

SUMMARY:
The purpose of this study is to investigate the effect of a family support program based on the nurse-led case management model on individuals providing care for patients who are confined to bed at home.

DETAILED DESCRIPTION:
It is of paramount importance to enable the patients receiving home care and their relatives to adapt social life, to fulfil their social integration, to relieve the burden of family members of the individual in need of care, especially the individual providing care, by supporting them in the environment where they live. In this study, it is aimed to investigate the effect of the family support program based on the nurse-led case management model for family members who care for bedridden patients.The family support program based on a five-stage nurse-led case management model is administered for the caregivers in the intervention group, the caregivers in the control group is monitored by home health services through routine follow-ups. The research will conducted as a randomized controlled study with an experimental design.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* To have been taking care of the caregiver for at least 6 months,
* Being literate
* Not to have sensory loss such as vision and hearing,
* Being open to communication and cooperation,
* Internet access and being able to use it,
* Having a phone where he can be reached,
* Not receiving any remuneration for the provision of care,
* Having a family bond with the person being cared for.

Exclusion Criteria:

* Caregivers who do not meet the inclusion criteria,
* Caregivers who did not give consent at any stage of the study and left.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Change in caregiver burden in 6 months | 6 months
  Zarit Caregiver Burden Scale: This scale was developed in 1980 by Zarit et al. to assess the stress experienced by those providing care to old people or to those in need of care. The lowest possible score is 0 and the highest is 88. A high score on the scale shows a high level of distress experienced.

SECONDARY OUTCOMES:
assessment of caregivers' quality of life | 6 months
  WHOQOL-BREF-TR Form: This form is the Turkish adaptation of the WHOQOL-100, which was developed by the World Health Organization to assess the quality of life of individuals. Cultural adaptation of the WHOQOL-BREF-TR in Turkey and validity and reliability work were conducted by Eser et al. (1999). This scale consists of 26 questions selected from the WHOQOL-BREF WHOQOL-100 scale. One item was added to the Turkish version of the scale.

OTHER OUTCOMES:
determination of family functional status | 6 months
  Family APGAR Scale: This scale, which evaluates the perceptions of family members concerning their functionality among themselves is used in determining the weak areas in family functions in a short time. The scale was developed by Smilkstein (1978) and adapted to Turkish in 2011 (Özcan et al. 2011). The Family APGAR Scale measures the five parameters of family functionality in adults of adaptation, partnership, growth, affection and resolve.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdanur Dikmen, Prof. Dr., Study Director — Sakarya University of Applied Sciences
Locations (1):
- Sakarya University of Applied Sciences, Sakarya, Turkey (Türkiye)